CLINICAL TRIAL: NCT02483754
Title: Application and Revision of Montreal Cognitive Assessment in Military Retirees With Mild Cognitive Impairment
Brief Title: Application and Revision of Montreal Cognitive Assessment in Chinese Retirees
Acronym: ARMOCA
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NCT02483754
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2015-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- original MOCA: The Chinese retired military cadres were surveyed with the revised MOCA scale.
- revised MOCA: The random part of participants were surveyed with the revised MOCA scale.

SUMMARY:
The study was designed to employ MOCA to screen mild cognitive impairment (MCI) in military retirees and to analyze the associated risk factors. As such, MOCA was revised to be validated for the Chinese context.

DETAILED DESCRIPTION:
Three hundred and four retired military cadres were investigated using a random cluster sampling technique including personal information, prevalence, MOCA scale, and related neuropsychiatry scale. Thirty retirees were random chosen and tested again with the revised MOCA scale one month later.

ELIGIBILITY:
Inclusion Criteria:

* aged >=60 years old retired military cadres lived in Xian,Shaanxi,China questionnaires completed

Exclusion Criteria:

* deaf-mute

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three hundred and four retired military cadres.They can be divided by age, level of education and physical exercise and cerebral apoplexy to evaluate their mild cognitive impairment.
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
MCI occurrence rate | up to 8 months
  Three hundred and four retired military cadres from 9 Xi'an military sanatoria were investigated，assessed up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Wang, Doctor, Study Chair — Air Force Military Medical University, China